CLINICAL TRIAL: NCT05978466
Title: MANAGEment of Atrial Fibrillation Outcomes Registry (MANAGE-AF)
Brief Title: MANAGE-AF Registry -MANAGEment of Atrial Fibrillation Outcomes Registry (MANAGE-AF)
Acronym: MANAGE-AF
Status: Recruiting | Type: Observational
Sponsor: CorVita Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-CSF-00100
Record Dates: First submitted 2019-04-11; First posted 2023-08-07 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial arrhythmia; atrial fibrillation; stroke; bleeding; Left Atrial Appendage Occlusion
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to learn more about the normal care of patients with a new or pre-existing diagnosis of atrial fibrillation (AF). These abnormal and irregular heartbeats place patients at increased risk of developing clots in their bloodstream that could potentially lead to stroke. Normal care is designed to help prevent this from happening and to lessen or eliminate the symptoms patients may have. There are many different types of AF as well as numerous ways in which a variety of patients are treated. The investigators are interested in gathering more information to better keep track of patient treatment patterns (trends) that may differ from physician to physician, hospital to hospital, medication to medication, patient to patient and if necessary, procedure to procedure.

DETAILED DESCRIPTION:
The objective of this research is to establish a contemporary and simple to construct AF management registry that expands progressively over the continuum of care for each individual patient. The registry will be used to determine the course and progression of AF management in preventing thrombo-embolic events using rhythm and rate control interventions.

Primary endpoints:

1. Atrial fibrillation natural history
2. Thrombo-embolic event
3. Death

Secondary endpoints:

1. Bleeding
2. Pro-arrhythmia
3. Patient adherence
4. Treatment complication

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of valvular or non valvular atrial fibrillation
2. ECG documented atrial fibrillation A. 12 lead B. Rhythm strip C. Event monitor D. Holter Monitor E. Implantable loop recorder

Exclusion Criteria:

1. Age below 18 years.
2. Clinical evidence that death within 6 months is possible
3. Inability to consent to the research or sign a consent form
4. Inability to follow up at the research clinic at least annually for continuity of AF care and management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects with the diagnosis of atrial fibrillation can be enrolled into the study regardless of sex, age or medical history
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Atrial fibrillation | From enrollment to 10- year study completion
  The natural progression of the condition will be assessed per medical record review
Number of participants who had thrombo-embolic event | From enrollment to 10- year study completion
  All strokes, transient ischemic and systemic thrombo-embolic events
Mortality | From enrollment to 10- year study completion
  All cause death will be noted

SECONDARY OUTCOMES:
Number of participants who have experienced bleeding | From enrollment to 10- year study completion
  All bleeding events events will be will be assessed throughout the duration of the study per medical record review
Number of patients who have had pro-arrhythmia events | From enrollment to 10- year study completion
  All pro-arrhythmic events will be documented and assessed
Number of patients who have had patient adherence events | From enrollment to 10- year study completion
  Events relating to subject non-compliance of medications will be documented for the duration of the study per medical record review
Treatment complication | From enrollment to 10- year study completion
  All adverse outcomes/events related to routine standard of care treatments will be noted and assessed for the duration of the study per medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Burke, DO, Principal Investigator — Chief Scientific Officer
Locations (1):
- CorVita Science Foundation (NFP), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish the results or outcomes associated with this registry to major peer-reviewed journals, didactic or poster sessions at national/international medical conferences.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Intermittently over the next 10-15 years
Access Criteria: Co-investigator who enrolls at least one patient
URL: http://www.corvitascience.org

REFERENCES:
- See also: Research foundation's website — http://www.corvitascience.org